CLINICAL TRIAL: NCT02508701
Title: A Pilot Study Comparing the Effectiveness of On-site Campus Interventions to Increase the Uptake of the HPV Three-shot Series Vaccine Among College Aged Men: A 2 X 2 Repeated Design
Brief Title: A Pilot Study Comparing the Effectiveness of Campus Intervention to Increase HPV Vaccine Rate Among College Aged Men
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Stewart Chang Alexander, Associate Professor, Purdue University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1506016224
Record Dates: First submitted 2015-07-24; First posted 2015-07-27 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Human Papilloma Virus, Male
Keywords: HPV; Message Design; Adolescent Males

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Altruistic inside-dorm (Other): Altruistic & personal message with direct recommendation and access to the vaccine on-site
  The intervention is a message asking students to get the vaccine that tell students the vaccine is available in the dorm and provides a direct recommendation to get the vaccine
  Interventions: Behavioral: Message X Onsite/Offsite Vaccination
- Generic inside-dorm (Other): Generic message and access to the vaccine on-site
  The intervention is a message asking students to get the vaccine that tell students the vaccine is available in the dorm but provides no recommendation
  Interventions: Behavioral: Message X Onsite/Offsite Vaccination
- Generic outside-dorm (Other): Generic message and off-site access to the vaccine
  The intervention is a message asking students to get the vaccine that tell students the vaccine is available at the health center but provides no recommendation
  Interventions: Behavioral: Message X Onsite/Offsite Vaccination
- Altruistic outside-dorm (Other): Altruistic & personal message with direct recommendation and off-site access to the vaccine
  The intervention is a message asking students to get the vaccine that tell students the vaccine is available at the student health center and provides a direct appeal to get the vaccine
  Interventions: Behavioral: Message X Onsite/Offsite Vaccination

INTERVENTIONS:
Behavioral: Message X Onsite/Offsite Vaccination — Personal, Altruistic Message vs Generic Message Inside-Dormitory Vaccination vs. Student Health Center Vaccination

SUMMARY:
This is a study testing what type of message and access influences a young male to get the HPV vaccine.

The investigators are conducting a 2 X 2 design

These conditions are:

* Condition 1: Altruistic personal with direct recommendation inside-dorm
* Condition 2: Generic message with inside-dorm
* Condition 3: Generic message with outside-dorm HPV vaccine
* Condition 4: Altruistic personal with outside-dorm HPV vaccine

The objectives of this study are:

A. To examine the efficacy in encouraging young men to receive HPV shots at Time 1 within each of the four intervention conditions (altruistic/personal with direct recommendation vs. generic message) X (in-dorm vs. outside-dorm HPV vaccine).

B. To examine the efficacy in encouraging young men to receive HPV shots at Times 2 & 3 within each of the four intervention conditions (altruistic/personal with direct recommendation vs. generic message) X (in-dorm vs. outside-dorm HPV vaccine).

2.1.1 List the clinical hypotheses. Objective A H A.1: At Time 1, college men who have immediate access to the HPV vaccination will take the vaccination at a higher rate than those who do not have immediate access to the vaccine.

H A.2: At Time 1, college men who receive an altruistic/personal health message along with immediate access to the HPV vaccine will take the HPV vaccination at a higher rate than the men in the other three arms of the study.

Objective B H B.1: At Times 2 & 3, college men who have immediate access to the HPV vaccination will take the vaccination at a higher rate than those who do not have immediate access to the vaccine.

H B.2: At Times 2 & 3, college men who receive an altruistic/personal health message along with immediate access to the HPV vaccine will take the HPV vaccination at a higher rate than the men in the other three arms of the study.

DETAILED DESCRIPTION:
The investigators will conduct an intervention on the Purdue campus targeting men-only dorm wings (living areas). Eight (8) dorm wings will be selected in advance.

Dorm wings will be randomly assigned to one of four intervention arms: (1) educational message with altruistic/personal health benefits emphasized along with a direct recommendation to get the vaccine along with immediate access to the vaccine with the dormitory (altruistic/personal benefit message with recommendation + in-dorm vaccine), (2) educational message with altruistic/personal health benefits emphasized along with information on where to go to get the vaccine (altruistic/personal benefit message with recommendation + outside-dorm vaccine) and (3) generic informational message about the HPV vaccine and immediate access to the vaccine in the dormitory (generic + on-site vaccine), (4) generic informational message with information on where to go to get the vaccine (generic + outside-dorm vaccine).

Phase 1 (Initial vaccine dose #1):

Recruitment of all four intervention arms will be occur at the same time during the dorm wing's first mandatory meetings for residents. These mandatory meetings occur throughout the campus. Fifty-two (52) residents live on each dorm wing and the first mandatory dorm meeting attendance is typically between 75-90% of all residents within the wing (between 47 and 52 men).

At the end of the mandatory wing meeting, a male research assistant will provide a brief presentation to the young men that describe the HPV vaccine (either altruistic/personal benefit message with recommendation or a generic message).

At the end of the brief presentation, residents will either be directed to the location where the HPV vaccine is set-up within the dormitory for immediate immunization (on-site vaccine) or provided a printed card that tells them how to get the vaccine on campus through the health center(outside-dorm vaccine). The location of the on-site vaccine will be close to the dorm wing.

Eligibility requirements will be determined at the site of the HPV vaccine by student health center staff members. These requirements are (over 18-years of age and have not received the three-shot series of the HPV vaccine).

For the on-site vaccine arms, once eligibility has been determined, research assistants will hand the young man over to the student health center staff (who will then conduct their typical vaccine protocol).

For those in the outside-dorm vaccine arms, students will go to the health center to receive the vaccine.

Phase 2 (2-month follow-up vaccine dose #2):

On-site vaccine arms. One week before the student health center staff will return to the dormitory for administer the second HPV dose, research assistants will contact participants by text and email to remind them of the follow-up. The investigators will also send a text message and email the night before. In addition, Resident Assistants will also be provided the name of the men in the study to remind participants of the returned visit the night before about the visit.

Outside-dorm vaccine. For those randomized to outside-dorm, research assistants will text and email participants one-week before their 2-month follow-up dose is needed. Resident Assistants will also be provided the name of the men in the study to remind participants about the getting the follow-up shot.

Phase 3: (6-month follow-up dose #3): The investigators will use the same protocol for the 6-month follow-up as the investigators use for the 2-month follow-up (reminder one week before and the night before using email, text, and resident assistants).

ELIGIBILITY:
Inclusion Criteria:

* Must be young men between 18 to 21 years old
* live in one of the dorm floors in the study

Exclusion Criteria:

* Under 17 years old
* over 21 years old
* females
* young men that live outside the pre-identified dorm halls
* Also any young man with a moderate to severe illness will be excluded.
* anyone with a life threatening allergic reaction to components to the HPV vaccine

Ages: 18 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart C Chang Alexander, PhD, Principal Investigator — Purdue University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Altruistic Inside-dorm: Altruistic & personal message with direct recommendation and access to the vaccine on-site
  Message X Onsite/Offsite Vaccination: Personal, Altruistic Message vs Generic Message Inside-Dormitory Vaccination vs. Student Health Center Vaccination
- Generic Inside-dorm: Generic message and access to the vaccine on-site
  Message X Onsite/Offsite Vaccination: Personal, Altruistic Message vs Generic Message Inside-Dormitory Vaccination vs. Student Health Center Vaccination
- Generic Outside-dorm: Generic message and off-site access to the vaccine
  Message X Onsite/Offsite Vaccination: Personal, Altruistic Message vs Generic Message Inside-Dormitory Vaccination vs. Student Health Center Vaccination
- Altruistic Outside-dorm: Altruistic & personal message with direct recommendation and off-site access to the vaccine
  Message X Onsite/Offsite Vaccination: Personal, Altruistic Message vs Generic Message Inside-Dormitory Vaccination vs. Student Health Center Vaccination
Period: Overall Study
Arm/Group | Altruistic Inside-dorm | Generic Inside-dorm | Generic Outside-dorm | Altruistic Outside-dorm
Started | 9 | 6 | 5 | 4
Completed | 0 | 1 | 0 | 1
Not Completed | 9 | 5 | 5 | 3
Not completed — Lost to Follow-up | 9 | 5 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Altruistic Inside-dorm | Generic Inside-dorm | Generic Outside-dorm | Altruistic Outside-dorm | Total
Number analyzed (Participants) | 9 | 6 | 5 | 4 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 5 | 4 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 9 | 6 | 5 | 4 | 24
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 5 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1st Uptake Shots
Description: Number of Participants with the 1st Uptake Shots
Time Frame: Up to 12 months
Population: Frequency
Measure: Number; unit: participants
Arm/Group | Altruistic Inside-dorm | Generic Inside-dorm | Generic Outside-dorm | Altruistic Outside-dorm
Number analyzed (Participants) | 9 | 6 | 5 | 4
participants | 9 | 6 | 5 | 4

2. Primary Outcome: Number of Participants With 1st Uptake Shot
Description: The Number of Participants with 1st Uptake Shot
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Altruistic Inside-dorm: Altruistic & personal message with direct recommendation and access to the vaccine on-site
  The intervention is a message asking students to get the vaccine that tell students the vaccine is available in the dorm and provides a direct recommendation to get the vaccine
  Message X Onsite/Offsite Vaccination: Personal, Altruistic Message vs Generic Message Inside-Dormitory Vaccination vs. Student Health Center Vaccination
- Generic Inside-dorm: Generic message and access to the vaccine on-site
  The intervention is a message asking students to get the vaccine that tell students the vaccine is available in the dorm but provides no recommendation
  Message X Onsite/Offsite Vaccination: Personal, Altruistic Message vs Generic Message Inside-Dormitory Vaccination vs. Student Health Center Vaccination
- Generic Outside-dorm: Generic message and off-site access to the vaccine
  The intervention is a message asking students to get the vaccine that tell students the vaccine is available at the health center but provides no recommendation
  Message X Onsite/Offsite Vaccination: Personal, Altruistic Message vs Generic Message Inside-Dormitory Vaccination vs. Student Health Center Vaccination
- Altruistic Outside-dorm: Altruistic & personal message with direct recommendation and off-site access to the vaccine
  The intervention is a message asking students to get the vaccine that tell students the vaccine is available at the student health center and provides a direct appeal to get the vaccine
  Message X Onsite/Offsite Vaccination: Personal, Altruistic Message vs Generic Message Inside-Dormitory Vaccination vs. Student Health Center Vaccination
Arm/Group | Altruistic Inside-dorm | Generic Inside-dorm | Generic Outside-dorm | Altruistic Outside-dorm
Number analyzed (Participants) | 9 | 6 | 5 | 4
Participants | 9 | 6 | 5 | 4

3. Secondary Outcome: Number of Participants With Second Uptake Shot
Time Frame: 6 months
Population: Data was not collected because study was terminated.
Arm/Group | Altruistic Inside-dorm | Generic Inside-dorm | Generic Outside-dorm | Altruistic Outside-dorm
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With 3rd Uptake Shots
Description: The Number of Participants with 3rd Uptake Shots
Time Frame: 6 months
Population: Study data on this outcome was not collected because study was terminated
Arm/Group | Altruistic Inside-dorm | Generic Inside-dorm | Generic Outside-dorm | Altruistic Outside-dorm
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Altruistic Inside-dorm | Generic Inside-dorm | Generic Outside-dorm | Altruistic Outside-dorm
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No